CLINICAL TRIAL: NCT03764904
Title: Airway Ultrasound as a Predictor for Postextubation Stridor in Cervical Spine Surgery [Anterior Approach]: Prospective Observational Study
Brief Title: Airway Ultrasound as a Predictor for Postextubation Stridor in Anterior Cervical Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Khairy Elbeialy, Lecturer of Anesthesia, Ain Shams University
Other Study IDs: FMASU R 68 /2018
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Postextubation Stridor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Airway Ultrasound — Laryngeal US will be performed with a 12 megahertz (MHz) linear probe attached to the ultrasound device. With the probe placed transversely on the midline of the anterior neck over the cricothyroid membrane.

SUMMARY:
literature on use of the ultrasound (US) in extubation decisions in cervical spine surgery is scarce.The aim of this study will be to evaluate the utility of US as an aid for decision making for extubation in elective cervical spine surgery (anterior approach) operations and as a predictor for postextubation stridor in these operations

ELIGIBILITY:
Inclusion Criteria:

* surgeries associated with either exposure of more than three vertebral bodies,
* exposures involving the C2-C4 levels,
* blood loss exceeding 300 mL
* surgical time of more than five hours,

Exclusion Criteria:

* laryngotracheobronchial pathology,
* severe cardiorespiratory disease,
* admitted for redo-surgery
* intubated prior to operation
* Patient with anesthetic risk factors include Mallampati 3 or 4 and multiple intubation attempts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Thirty patients aged 18-60 years ASA Ⅰ and Ⅱ of both genders who are scheduled for elective anterior cervical surgery under general anesthesia in supine position for the first time will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the correlation between the post procedural laryngeal air-column width difference [LACWD] as obtained by laryngeal US with occurrence of postextubation stridor | First 6 hours postoperatively
  At the end of operation, laryngeal air column width [which is defined as the width of air between the vocal cords as demonstrated by US] will be obtained while the tube cuff is inflated then while it is deflated for three consecutive respiratory cycles after gentle suction of oropharyngeal airway. The laryngeal air-column width difference [LACWD] (the difference between width at balloon-cuff deflation and at balloon-cuff inflation) will be obtained and the average value will be recorded.
  Patient will be considered ready for extubation after performance of the cuff-leak test as [the volume of reduced cuff leak test is more than 110 ml] then reversal of neuromuscular blockade will be done. They tube will be removed when the patients can open their eyes on verbal commands and the T4/T1 ratio is 90% or more.
  After transferal of patients ICU where they will be observed for occurrence of postextubation stridor in the first 6 hour postoperatively.

SECONDARY OUTCOMES:
Incidence of other airway complication as hematoma | Intraoperative pre-extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided